CLINICAL TRIAL: NCT02906943
Title: Ontario-wide Cancer TArgeted Nucleic Acid Evaluation
Acronym: OCTANE
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: OCTANE
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Lung Cancer; Colorectal Cancer; Melanoma; Gynecological Cancer; Genitourinary Cancer; Pancreatobiliary Cancer; Gastrointestinal Cancer; Head and Neck Cancer; Rare Cancer; Unknown Primary Cancer
Keywords: Molecular Profiling; Advanced Cancer; Advanced Solid Tumors; Phase I Clinical Trial Candidates; Next Generation Sequencing
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Melanoma; Urogenital Neoplasms; Gastrointestinal Neoplasms; Head and Neck Neoplasms; Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tumor tissue 2 tubes of whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced cancer: Patients with advanced, incurable solid tumors receiving standard palliative treatment(s) will have archival tumor specimens requested and used for targeted next generation sequencing (NGS) testing. Blood samples and additional archival tumor specimens will be collected for banking and future research purposes.

SUMMARY:
Substantial progress has been made in the treatment of cancer through the use of targeted therapies, but what works for one patient might not work for another patient. Certain drugs are now being developed that target specific molecules in the body that are believed to be part of the disease.

Biomarkers are specific characteristics of the cancer that may help provide prognostic information (e.g. how well patients will be regardless of the treatments given) or help predict sensitivity or resistance to a specific treatment.

The study will collect archival tumor samples (previously collected biopsy or surgical tumor samples) to provide biomarker data about a patient's cancer, which may help their physicians to identify which clinical trials of new drug treatments may be most appropriate for the patient in the future and may also guide the use of approved treatments that may potentially benefit the patient.

Another goal of this study is to develop a province-wide registry of targeted gene sequencing testing results that will be made available to cancer researchers. Additional tumour tissue and blood samples collected from all study participants will also be stored in a biobank at the Ontario Institute for Cancer Research for future research.

The study will also look at linking data from this study to other health care databases to further collect information about the health care the patients received, including medical tests, clinic visits, or procedures both before and after participating in this study. Having more information about patient health to relate to the DNA sequences may provide new insights into cancer and its treatment.

DETAILED DESCRIPTION:
A recent survey of clinical genetic testing laboratories for cancer diagnostics by the Molecular Oncology Advisory Committee for Cancer Care Ontario identified disparities in access and use patterns for next generation sequencing (NGS) across the province of Ontario. All fourteen responding laboratories indicated that NGS instruments were either currently being used for clinical testing, were in the validation stage, or that they were planning to purchase NGS instruments within the near future. Respondents were uncertain about what tests should be performed, how costing and reimbursement would be addressed by the provincial funding agency (e.g. individual tests vs. panels), and how to deal with informatics issues from NGS testing, such as storage, variant interpretation, and utilization over the long term.

Given the increasing use of multi-gene somatic mutation testing in routine clinical cancer care (e.g. KRAS, NRAS, BRAF mutations in colorectal cancer, EGFR mutation and ALK translocation in non-small cell lung cancer, and BRAF, NRAS, and cKIT mutations in malignant melanoma), there is a need to expand the infrastructure for NGS panel testing in clinical laboratories. With a single payer provincial health care system, there is also an opportunity to develop a provincial-wide registry of NGS panel-based testing results and repository of genomically-characterized and clinically-annotated tumor tissues and blood samples to accelerate the development of additional "omic"-based tests for clinical use.

This study will enroll patients with advanced, incurable solid tumors at selected Ontario hospitals receiving standard palliative treatment(s). Archival formalin-fixed paraffin embedded (FFPE) tumor tissue will be requested and undergo targeted panel sequencing. An additional FFPE tissue sample will be requested at the same time for future research purposes. Patients will also be asked to provide blood samples for future research. A selected number of genes will be annotated in a research report provided to their treating oncologist. In addition to the clinically reported variants, targeted NGS testing results for all tested genes will be captured in a clinical research database that can be accessed by the treating oncologist in a secure web-based portal.

Following the reporting of targeted DNA sequencing results into the web-portal, remaining tumor DNA will be stored in the clinical testing laboratories. Blood samples collected at the time of consent and additional FFPE research blocks or slides collected for research will be transferred to a centralized biorepository maintained by the Ontario Tumour Bank (OTB) for more comprehensive analysis at the Princess Margaret (PM)-Ontario Institute for Cancer Research (OICR) Translational Genomics Laboratory (TGL). Blood will undergo standard germline DNA extraction and plasma processing for future circulating tumor DNA (ctDNA) and RNA (ctRNA) isolation at the PM-OICR TGL. Selected patient samples will be further characterized at the PM-OICR TGL for test development, additional sequencing, or discovery research.

All patients will be asked to provide permission for data-sharing with other cancer researchers. The consent will also include a provision for review of patient health records through review of patient charts or administrative databases (i.e. Cancer Care Ontario New Drug Funding Program, Provincial Cancer Registry, etc.) to obtain addition information about time on drug treatments and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmation of advanced solid tumor malignancies who are candidates for systemic therapy.
2. All patients must have sufficient FFPE archived tumor tissue for molecular profiling.
3. Patient must be ≥ 18 years old.
4. Patient's ECOG performance status equal to 0 or 1.
5. All patients must have a life expectancy of > 6 months.
6. All patients must have adequate organ functions.
7. All patients must have signed and dated an informed consent form.

Exclusion Criteria:

1. Patients must not have received more than 2 lines of prior cytotoxic therapy for their recurrent/metastatic disease, with the exception of Phase I trial candidates who will not be excluded if more than 2 lines of prior cytotoxic therapy have been received.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced solid tumor malignancies, where archived formalin-fixed paraffin embedded (FFPE) is available and adequate for molecular profiling.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients included in a province-wide registry of NGS panel-based testing results | 5 years
Change in use of NGS panel-based testing in Ontario clinical genetic testing laboratories | 5 years
Number of patients included in province-wide repository of genomically-characterized tumour tissue and blood samples and their utilization rates for future research | 5 years
Change in rates of genomics based clinical research in Ontario | 5 years
Utilization rates of province-wide genomically-characterized and clinically-annotated patient base in enrollment into specific research initiatives | 5 years
Utilization rates of molecular profiling information provided to treating physicians in guiding future treatment decisions | 5 years

SECONDARY OUTCOMES:
Percentage of successful linkages between transferred study data and administrative databases | 5 years
Concordance between administrative data and clinically abstracted data comparing variables using 2x2 concordance tables | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, MD, Principal Investigator — Princess Margaret Hospital, Canada; Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (7):
- Canada (7):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Targeted gene sequencing results, along with limited clinical information that does not identify the patient as an individual, such as age, partial date of birth (year, month), gender, cancer type, and pathology information related to the samples tested, and survival time will be sent to centralized scientific databases or shared with collaborating researchers.
  Data from this study can be shared through two types of databases: open-access or controlled-access. An open-access database is publicly accessible and contains limited clinical information and analyses of samples. A controlled-access database contains more detailed clinical information, such as relevant past medical history and the results of prior and ongoing cancer treatments, and analyses of samples, but is only accessible to researchers who sign agreements defining how data may be used. All data will be stripped of all personal identifying information.

REFERENCES:
- [Derived] Kappel C, Jiang DM, Wong B, Zhang T, Selvarajah S, Warner E, Hansen AR, Fallah-Rad N, Sacher AG, Stockley TL, Bedard PL, Sridhar SS. Comprehensive genomic profiling of treatment resistant metastatic castrate sensitive prostate cancer reveals high frequency of potential therapeutic targets. Clin Genitourin Cancer. 2022 Jun;20(3):278-284. doi: 10.1016/j.clgc.2022.02.004. Epub 2022 Feb 22. PMID 35337750
- [Derived] Ma LX, Espin-Garcia O, Bedard PL, Stockley T, Prince R, Mete O, Krzyzanowska MK. Clinical Application of Next-Generation Sequencing in Advanced Thyroid Cancers. Thyroid. 2022 Jun;32(6):657-666. doi: 10.1089/thy.2021.0542. Epub 2022 May 16. PMID 35262412